CLINICAL TRIAL: NCT06058845
Title: Efficacy of Tamarindus Indica Fruit Juice in Optimizing Cardiometabolic Health of Patients Living With HIV and Elevated Triglycerides
Brief Title: Efficacy of Tamarindus Indica Fruit Juice in Optimizing Cardiometabolic Health of Patients Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Mildmay Uganda Limited (Other)
Responsible Party: Principal Investigator, Christophe Matthys, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tamarind_001
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cardiometabolic Syndrome; Dyslipidemias; Hypertension
Keywords: Vascular function; Tamarindus indica; Lipid metabolism; Glucose metabolism; Polyphenols; HIV
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias; Hypertension

STUDY DESIGN:
Intervention Model Description: This is a single centre, 2-arm, 4 weeks randomised, double-blinded parallel trial with equal allocation ratios (1:1)
Who Masked: Participant, Investigator
Masking Description: Both participants and the study team will be blinded to the intervention materials. The two juice prototypes will be blinded by assigning a secret code to each of the intervention products. As such, blinding of the investigators and participants will be undertaken to ensure a double-blind intervention. Moreover, the statistical analyses of the main endpoints will be done before breaking the intervention product concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10% Tamarindus indica fruit pulp juice (Active Comparator): Participants will follow a daily consumption of 600ml of Tamarindus indica fruit juice containing 10% Tamarindus indica fruit pulp for 30 days
  Interventions: Dietary Supplement: Tamarindus indica fruit juice_A
- 30% Tamarindus indica fruit pulp juice (Experimental): Participants will follow a daily consumption of 600ml of Tamarindus indica fruit juice containing 30% Tamarindus indica fruit pulp for 30 days
  Interventions: Dietary Supplement: Tamarindus indica fruit juice_B

INTERVENTIONS:
Dietary Supplement: Tamarindus indica fruit juice_A — The participants will be exposed to 10% Tamarind pulp juice
  Arms: 10% Tamarindus indica fruit pulp juice
Dietary Supplement: Tamarindus indica fruit juice_B — The participants will be exposed to 30% Tamarind pulp juice
  Arms: 30% Tamarindus indica fruit pulp juice

SUMMARY:
The increasing burden of metabolic disturbances among People Living with HIV especially in developing countries has posed need for scientifically-proven, innovative, sustainable and cost-effective local adjuvant remedies to supplement conventional medical interventions. The goal of this clinical trial is to test the potential of Tamarindus indica fruit juice to improve cardiometabolic health of PLWH and elevated Triglycerides (TG). The main aims it aims to answer are to;

* evaluate the efficacy of T. indica fruit juice on selected markers of lipid and glucose metabolism, and vascular health.
* investigate a possible dose-response relationship on cardiometabolic control following intake of varying concentrations (fruit pulp percentages) of T. indica fruit juice.

Participants will be required to consume 600 ml of either 10% or 30% fruit pulp juice a day for 30 days. From the baseline measurements, participants will be asked to comeback for repeat measurements after 14 days and finally on the 3oth day (Endline). Researchers will compare the groups that will be expose to the two juice prototypes to determine potential differences in TG levels.

DETAILED DESCRIPTION:
Suboptimal cardiometabolic health is on a disproportional rise in Low- and Middle-Income Countries (LMICs). In sub-Saharan Africa (SSA), cardiometabolic dysfunction is being exacerbated by the ongoing nutrition transition, that has seen a change from traditional diets to fast and ultra processed foods rich in sugar, fats, and salt coupled by low physical activity (Kiyimba et al., 2022). Similarly, chronic inflammatory diseases such as HIV can aggravate cardiometabolic risks (Todowedo et al., 2019). Beyond conventional nutrients, fruits and vegetables have ubiquitous amounts of bioactive components including polyphenols, alkaloids, saponins, and terpenes and terpenoids, with polyphenols being the most ubiquitous of all. Dietary polyphenols are a diverse category of secondary plant metabolites that represent the largest group of naturally occurring antioxidants with cardioprotective benefits (Rijha et al., 2022 and Quero et al., 2020). Our recent inventory study of Uganda's IFV with purported cardiometabolic benefits, highlighted the popularity of Tamarindus indica as a local adjuvant therapy for cardiometabolic risks among Ugandan communities (Kiyimba et al., 2023).

T. indica, is a leguminous tree belonging to the family Fabaceae with a wide range of bioactive constituents in varying levels- the highest being polyphenols followed by alkaloids, saponins, and terpenoids in that order (Luca et al., 2019 and Penev et al., 2016). Therefore, the aim of this trial is to evaluate the efficacy of T. indica fruit juice (added to patients' usual diets) on selected cardiometabolic risk markers of PLWH under the community-based HIV care model in Uganda in a proof-of-concept clinical trial. Two blinded juice prototypes of 10% and 30% fruit pulp packaged in amber bottles each consisting of 300mls will be supplied by the Uganda Natural Chemotherapeutics Research Institute.

This is a single centre, 2-arm, 4 weeks randomised, double-blinded parallel trial with equal allocation ratios. The study participants will be randomly allocated to consume twice-daily 600 mL of either 10% or 30% pulp of T. indica fruit juice. Both participants and the study team will be blinded to the intervention materials. Measurements will be performed at three different timelines: Baseline, Week two of the study, and Endline (week four of the study). Compliance to the study protocol will be confirmed by weekly telephone inquiries, and by counting the returned empty juice bottles or unused study products at each follow-up visit. Participants will be asked to maintain their habitual dietary regimen. The two juice prototypes will be blinded by assigning a secret code to each of the intervention products. As such, blinding of the investigators and participants will be undertaken to ensure a double-blind intervention. Moreover, the statistical analyses of the main endpoints will be done before breaking the intervention product concealment.

ELIGIBILITY:
Inclusion Criteria:

* Triglycerides ≥150 mg/dL
* TLD regimen (ART) for ≥12 months
* 95% ART adherence in last 6 months
* Virally suppressed (most recent results viral load suppressed within the last 12 months)
* PLWH aged ≥30≤60 years.
* No plans to change location in the next 6 months

Exclusion Criteria:

* Taking dietary supplements
* TB co-infection, renal failure disease, liver cirrhosis, chronic pancreatitis
* Pregnancy and Lactation or regular sport activity
* Parallel participation in another clinical trial
* On treatment for; dyslipidemia, hypertension or diabetes and oral hypoglycemic drugs
* Very low blood pressure (< 90/50 mmHg)
* Not willing to consent or unable to consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in the concentrations of Triglycerides | 30 days
  A 10 mg/dL reduction in plasma triglycerides

SECONDARY OUTCOMES:
Changes in the concentrations of Total cholesterol | 30 days
  Reduction in plasma cholesterol
Changes in the concentrations of LDL-c | 30 days
  Reduction in plasma LDL-c
Changes in the concentration of HDL-c | 30 days
  increase in plasma HDL-c
Changes in the concentrations of Fasting Blood Glucose (FBG) | 30 days
  Reduction in FBG
Changes in Pulse wave velocity (m/s) | 30 days
  Measure of arterial stiffness (improvement in vascular function)
Changes in mmHg of Blood pressure | 30 days
  Improvement in both systolic and diastolic blood pressure

OTHER OUTCOMES:
Changes in Waist circumference (WC) | 30 days
  Reduction in WC
Changes in Kg of body's fat mass | 30 days
  Improvement in fat mass (reduction)
Changes in Body weight | 30 days
  reduction in body weight
Changes in BMI | 30 days
  reduction in BMI

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Matthys, PhD, Study Director — KU Leuven
Locations (1):
- Kajjansi HCIV, Wakiso, Uganda

IPD SHARING:
Plan to Share IPD: Yes
For all the data generated during the course of this study, we will follow the prevailing standards and guidelines in documenting and depositing data sets.
  The research team will disseminate results from this research through presentations at public lectures, scientific institutions and meetings, and/or publication in major journals. Regarding data sharing, International Committee of Medical Journal Editors recommendations will be followed.
  Individual deidentified participant data will be shared. In particular, individual participant data that underlie the results reported in our articles, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will become available from 9-36 months after the publication of the study-results by the research team.
Access Criteria: Data will only be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals should be directed to Prof. Christophe Matthys (Christophe.matthys@uzleuven.be). To gain access, data requestors will need to sign a data access agreement

REFERENCES:
- [Background] Todowede OO, Mianda SZ, Sartorius B. Prevalence of metabolic syndrome among HIV-positive and HIV-negative populations in sub-Saharan Africa-a systematic review and meta-analysis. Syst Rev. 2019 Jan 3;8(1):4. doi: 10.1186/s13643-018-0927-y. PMID 30606249
- [Background] Kiyimba T, Kigozi F, Yiga P, Mukasa B, Ogwok P, Van der Schueren B, Matthys C. The cardiometabolic profile and related dietary intake of Ugandans living with HIV and AIDS. Front Nutr. 2022 Aug 11;9:976744. doi: 10.3389/fnut.2022.976744. eCollection 2022. PMID 36034927
- [Background] Rajha HN, Paule A, Aragones G, Barbosa M, Caddeo C, Debs E, Dinkova R, Eckert GP, Fontana A, Gebrayel P, Maroun RG, Napolitano A, Panzella L, Pasinetti GM, Stevens JF, Schieber A, Edeas M. Recent Advances in Research on Polyphenols: Effects on Microbiota, Metabolism, and Health. Mol Nutr Food Res. 2022 Jan;66(1):e2100670. doi: 10.1002/mnfr.202100670. Epub 2021 Dec 2. PMID 34806294
- [Background] Quero J, Marmol I, Cerrada E, Rodriguez-Yoldi MJ. Insight into the potential application of polyphenol-rich dietary intervention in degenerative disease management. Food Funct. 2020 Apr 30;11(4):2805-2825. doi: 10.1039/d0fo00216j. PMID 32134090
- [Background] Luca SV, Macovei I, Bujor A, Miron A, Skalicka-Wozniak K, Aprotosoaie AC, Trifan A. Bioactivity of dietary polyphenols: The role of metabolites. Crit Rev Food Sci Nutr. 2020;60(4):626-659. doi: 10.1080/10408398.2018.1546669. Epub 2019 Jan 7. PMID 30614249
- [Background] Penev L, Paton A, Nicolson N, Kirk P, Pyle RL, Whitton R, Georgiev T, Barker C, Hopkins C, Robert V, Biserkov J, Stoev P. A common registration-to-publication automated pipeline for nomenclatural acts for higher plants (International Plant Names Index, IPNI), fungi (Index Fungorum, MycoBank) and animals (ZooBank). Zookeys. 2016 Jan 7;(550):233-46. doi: 10.3897/zookeys.550.9551. eCollection 2016. PMID 26877662

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT06058845/Prot_SAP_000.pdf